CLINICAL TRIAL: NCT01628575
Title: Periodontally Accelerated Orthodontics - A Novel Technique For a Shortened Orthodontic Treatment With a Stable Result. A Clinical and Computerized Tomography Analysis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Tali Chackartchi, DMD, Hadassah Medical Organization
Other Study IDs: HMO-0626-11
Record Dates: First submitted 2012-06-23; First posted 2012-06-27 (Estimated); Last update posted 2012-06-27 (Estimated); Status verified 2012-06

CONDITIONS: Periodontal Status of Patients Treated With PAO Tec
Keywords: periodontally accelerated orthodontics PAO

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- PAO: patients undergoing orthodontic treatment with the addition of pretreatment periodontal surgery for bone decortication.
  Interventions: Procedure: PAO

INTERVENTIONS:
Procedure: PAO — all patients underwent periodontal surgery for bone decortication followed by orthodontic treatment

SUMMARY:
Periodontally accelerated orthodontics, also known as PAO, is a novel technique combining alveolar corticotomy and bone grafting prior to commencing orthodontic treatment. Using this technique orthodontic de-crowding and space closing, can be completed in 60-70% less active orthodontic treatment time. The addition of particulated bone graft following decortication allows for the widening of the bucco-lingual alveolar bony dimension, thus creating space for the movement of teeth, without the creation of dehiscences, usually a negative sequel of the standard orthodontic treatment.

Aim: To evaluate the use of the PAO technique for the treatment of 20 adult patients 1 year post orthodontic treatment.

Methods: 20 periodontally healthy adult patients requiring orthodontic treatment were admitted in the departments of Periodontics and Orthodontics in Hadassah Medical Center. All patients underwent full orthodontic and periodontal examination upon admission including a pretreatment CBCT scan. Decortication followed by grafting was made after the orthodontic appliances have been placed. The orthodontic appliances were activated immediately after surgery and every 2 weeks. During the 1 year follow up a periodontal and orthodontic clinical evaluation were made, as well as a CBCT scan.

DETAILED DESCRIPTION:
20 patients were periodontally and orthodontically examined. including: full chart:ppd, free gin line, bleeding on probing, plaque score, teeth mobility. cephalometric analysis, clinical photographes, full periapical x rays.

perio=ortho treatment plan was scheduled, a periodontal surgery for the decortication of buccal bone and bone grafting was preformed.

at the same day orthodontic appliances were activated. in the follow up exam a full periodontal exam will be made (as at the beginning).

the patient will be referred to CBCT scan. all dicom files will be uploaded to simplant software, and measurements will be made: buccal bone width from crest to apex. distance from CEJ to crest. presence of root dehiscence and fenestrations. root resorption.

clinical measurements:

* recessions
* vas

ELIGIBILITY:
Inclusion Criteria:

* orthodontic treatment with periodontal surgery

Exclusion Criteria:

* smoking alcohol consumption pregnancy

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients from the department of orthodontics Hadassah medical center
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2012-12 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
buccal bone width | 1 year

SECONDARY OUTCOMES:
recessions | 1 year
  location of free gingival margin acording to CEJ
root resorption | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tali Chackartchi, DMD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Department of periodontology, Jerusalem, Israel